CLINICAL TRIAL: NCT07126210
Title: Peking University-Family Engaged, Enhanced Diet, for Kids (PKU-FeeD)
Brief Title: Weight Management Program for Obese Preschool Children
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Peking University (Other)
Collaborators: Shandong Maternal and Child Health Hospital (Unknown)
Responsible Party: Principal Investigator, Hai-Jun Wang, Professor in Department of Maternal and Child Health, School of Public Health, Peking University, Peking University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: IRB00001052-25071
Record Dates: First submitted 2025-08-01; First posted 2025-08-17 (Actual); Last update posted 2025-08-17 (Actual); Status verified 2025-08

CONDITIONS: Childhood Obesity
Keywords: Obesity; Intervention; Preschool; Management; Children
MeSH Terms: conditions — Pediatric Obesity; Obesity

STUDY DESIGN:
Who Masked: Outcomes Assessor
Masking Description: Randomization will be performed after the baseline survey. The assessors measuring childrens' health indicators will be blinded at follow-up phases.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- multicomponent intervention (Experimental): This study adopts a multicomponent intervention based on the "3 Less, 2 More, 1 Team" approach-Less fried/fatty foods, less sugar, less overeating; More colorful foods, more physical activity; and One team (family working together to raise a healthy child). The intervention is family-centered, supported by kindergartens and hospitals, with digital health technology.
  Interventions: Behavioral: Family engaged, enhanced Diet intervention
- usual-care control (No Intervention): In the control group, participating preschools will receive no intervention during the study period and will continue their routine educational and management practices without modification. After the study is fully completed, control group preschools will receive access to all intervention materials and health education resources developed for this project.

INTERVENTIONS:
Behavioral: Family engaged, enhanced Diet intervention — The family component includes health education via books, lectures, and short videos, parenting skills training, regular monitoring of child growth, and behavior goal setting through the mobile health platform. Motivational interviewing via telephone provides tailored behavioral support.
  Kindergartens assist in health education, supervise dietary intake and physical activity, monitor children's growth monthly, and maintain communication with families.
  Hospitals provide targeted health counseling and facilitate clinic access as needed.
  The mobile health platform integrates modules for health education, smart growth curve tracking, behavior goal management, and home-school-hospital collaboration.
  Arms: multicomponent intervention

SUMMARY:
The PKU-FeeD trial is a cluster-randomized controlled trial conducted in Jinan, Shandong Province, China. This study aims to: 1) Develop and evaluate a digital health-assisted, multidisciplinary intervention for preschool children with obesity, assessing its effectiveness and cost-effectiveness. 2) Investigate how lifestyle-based interventions influence the composition and function of the gut microbiota in obese preschoolers, and elucidate the mechanisms by which these interventions may modulate gut microbiota to affect obesity-related metabolic phenotypes.

DETAILED DESCRIPTION:
Childhood obesity has become a global public health challenge, and early prevention and management are crucial to curbing its epidemic. However, compared to school-aged children, evidence on effective obesity interventions for preschoolers remains limited and inconsistent. While preventive approaches may have broader population-level implications, targeted management interventions may be more cost-effective in settings with lower obesity prevalence but rising trends, providing foundational evidence for future preventive strategies.

The gut microbiota plays a key role in host energy metabolism and metabolic homeostasis, and its dysbiosis is strongly linked to obesity. Diet and physical activity, as core components of lifestyle interventions, may significantly shape gut microbial ecology, potentially influencing host metabolism and obesity-related outcomes. However, due to challenges in sample collection, existing studies on gut microbiota in children are scarce, with small sample sizes, and few intervention studies have established causal relationships. The interplay between healthy lifestyle interventions, gut microbiota, and childhood obesity remains understudied, and the underlying mechanisms require further exploration. Thus, this trial seeks to: 1) determine effectiveness of a digital health-supported, comprehensive intervention for preschool obesity management. 2) Elucidate causal relationships between dietary behaviors, gut microbiota, and obesity in preschoolers.

ELIGIBILITY:
Inclusion Criteria:

* The child's primary caregivers can proficiently use smart phones.
* Child is expected to remain in the same kindergarten for at least one year.
* No use of antibiotics or probiotic supplements, no acute stress events (e.g., trauma or severe infection), gastrointestinal symptoms (e.g., abdominal pain, constipation, diarrhea), or vaccinations within the 3 months prior to stool sample collection.
* Parents voluntarily agree to participate in the study and provide written informed consent.

Exclusion Criteria:

* Obesity caused by genetic factors, diseases (e.g., endocrine disorders, central nervous system damage), or medication use.
* History of major organ diseases, including cardiovascular, pulmonary, hepatic, or renal conditions (e.g., heart disease, hypertension, asthma).
* Children following special diets (e.g., vegetarians).
* Children with pathological eating disorders or medical conditions that limit physical activity.

Ages: 4 Years to 6 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 200 (Estimated)
Dates: Start 2025-09-15 (Estimated); Primary Completion 2026-06-30 (Estimated); Study Completion 2027-06-30 (Estimated)

PRIMARY OUTCOMES:
children's BMI-Z change | at end of the 9-month intervention
  Calculated based on height and weight using WHO standards. The primary outcome is the difference between two arms in the change of children's BMI-Z scores from baseline to the end of the intervention.

SECONDARY OUTCOMES:
children's BMI-Z change | at 21-month follow-up.
  Calculated based on height and weight using WHO standards. The primary outcome is the difference between two arms in the change of children's BMI-Z scores from baseline to follow-up.
Body Mass Index (BMI) | at the end of the 9-month intervention; at 21-month follow-up.
  BMI is calculated from measured height and weight.
Waist Circumference | at the end of the 9-month intervention; at 21-month follow-up
  Waist circumference is measured at the midpoint between the lower margin of the last palpable rib and the top of the iliac crest to evaluate central adiposity.
waist-to-Height Ratio, WHtR | at the end of the 9-month intervention; at 21-month follow-up.
  Calculated by dividing waist circumference by height, used as an indicator of fat distribution and risk for metabolic complications.
Systolic and Diastolic Blood Pressures | at the end of the 9-month intervention; at 21-month follow-up.
  Blood pressure is measured using an electronic sphygmomanometer with the child seated after resting, to assess cardiovascular health.
Body Composition | at the end of the 9-month intervention
  Body fat percentage is assessed using a bioelectrical impedance analyzer (MC-780A, TANITA, Tokyo, Japan).
Prevalence and Incidence of Overweight/Obesity | at the end of the 9-month intervention; at 21-month follow-up
  The proportion of children classified as overweight or obese according to WHO and Chinese standards, including newly identified cases at follow-up.
Dietary Intake | at the end of the 9-month intervention
  Total energy intake, macronutrient distribution, and food group consumption will be assessed using three consecutive 24-hour dietary recalls. Changes in dietary quality and structure will be evaluated.
Children's Eating Behaviors | at the end of the 9-month intervention
  Assessed using the Children's Eating Behavior Questionnaire (CEBQ), measuring dimensions such as food responsiveness, satiety responsiveness, and emotional eating
Parental Feeding Practices (CPCFBS) | at the end of the 9-month intervention
  Measured using the Chinese Preschooler's Caregivers Feeding Behavior Scale (CPCFBS), evaluating dimensions such as monitoring, pressure to eat, and food restriction.
Time Spent in Physical Activity | at the end of the 9-month intervention
  1)Children will wear an ActiGraph accelerometer for 7 consecutive days. Time spent in light, moderate, and vigorous physical activity will be calculated to evaluate changes in physical activity patterns. 2) Evaluated using the Children's Leisure Activities Study Survey (CLASS), assessing the amount and type of physical activity and sedentary behavior, including screen time.
Sedentary Behavior and Screen Time | at the end of the 9-month intervention
  1)Children will wear an ActiGraph accelerometer for 7 consecutive days. Time spent in light, moderate, and vigorous physical activity will be calculated to evaluate changes in physical activity patterns. 2) Evaluated using the Children's Leisure Activities Study Survey (CLASS), assessing the amount and type of physical activity and sedentary behavior, including screen time.
Gut Microbial Composition | at the end of the 9-month intervention
  Stool samples will be collected at baseline and post-intervention. Gut microbial composition is measured by 16S rRNA sequencing

CONTACTS AND LOCATIONS:
Overall Officials: Haijun Wang, PhD, Principal Investigator — Peking University
Locations (1):
- Department of Maternal and Child Health, School of Public Health, Beijing, Beijing Municipality, China

IPD SHARING:
Plan to Share IPD: No
Individual participant data (IPD) will not be shared publicly due to ethical considerations. In accordance with the study's ethical approval and informed consent procedures, the data contain potentially sensitive personal health information and are protected to ensure participant confidentiality and privacy. Data access is therefore restricted to authorized research personnel only and cannot be made publicly available.